CLINICAL TRIAL: NCT02290431
Title: A Phase II, Multi-center, Single Arm, Open Label Study to Evaluate the Efficacy and Safety of Panobinostat in Combination With Bortezomib and Dexamethasone in Japanese Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Panobinostat in Combination With Bortezomib and Dexamethasone in Japanese Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589D1201
Record Dates: First submitted 2014-10-24; First posted 2014-11-14 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Relapse/Refractory Multiple Myeloma
Keywords: LBH589; panobinostat; bortezomib; dexamethasone; Phase II; bortezomib and dexamethasone; Japanese patients; relapsed/refractory multiple myeloma; Panobinostat (PAN)
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Panobinostat; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBH589 + bortezomib + dexamethasone (Experimental): Participants were administered LBH589 (panobinostat)in combination with bortezomib and dexamethasone 2 weeks on/1 week off.
  Interventions: Drug: LBH589 (panobinostat); Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: LBH589 (panobinostat) — Panobinostat (PAN) capsules were supplied at dose strengths of 10 mg and 15 mg. and dosed at 20mg during treatment phase 1 (21 days) and treatment phase 2 (42 days)
Drug: bortezomib — Bortezomib (BTZ) s.c: 1.3 mg/m2 was administered during both treatment phase 1 (21 days) & treatment phase 2 (42 days).
Drug: dexamethasone — Dexamethasone (Dex): 20mg tablets taken during both treatment phase 1 (21 days & treatment phase 2 (42 days)

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of panobinostat in combination with bortezomib and dexamethasone in Japanese patients with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient had a previous diagnosis of multiple myeloma
* Patient required retreatment for multiple myeloma
* Patient had measurable M component in serum or urine at study screening

Exclusion Criteria:

* Primary refractory disease (patients that never reached at least an minor response for over 60 days under any prior therapy)
* Patient who had been treated by bortezomib before, and did not reach at least a minor response under this therapy, or progressed under it or within 60 days of last dose
* Patient received prior treatment with DAC inhibitors including panobinostat
* Patient had impaired cardiac function, or a prolonged QTc interval at screening ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Japan (20):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Shibukawa, Gunma
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Tokushima

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Suzuki K, Sunami K, Matsumoto M, Maki A, Shimada F, Suzuki K, Shimizu K. Phase II, Multicenter, Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of Panobinostat in Combination with Bortezomib and Dexamethasone in Japanese Patients with Relapsed or Relapsed-and-Refractory Multiple Myeloma. Acta Haematol. 2021;144(3):264-274. doi: 10.1159/000508529. Epub 2020 Dec 4. PMID 33279887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 33 eligible subjects were planned to be enrolled. 31 eligible subjects were enrolled and treated with PAN+BTZ+Dex (Treatment phase 1), of which 17 subjects entered Treatment phase 2. All 31 subjects entered the post-treatment evaluation phase, of which 22 discontinued the study. 24 subjects entered the survival follow-up phase.
Period: Overall Study
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Started | 31
Subjects. Discont. Prematurely | 27
Subjects Completed Study Per Protocol | 8
Subjs. Ntered Post-treatment Eval. Phase | 31
Subjects Entered Survival f/u Phase | 24
Entered Treatment Phase 2 | 17
Completed | 4
Not Completed | 27
Not completed — Adverse Event | 20
Not completed — Progressive disease | 4
Not completed — Study terminated by Sponsor | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) comprised of all subjects who took at least one dose of any study treatment component.
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Near Complete Response (nCR)/ Complete Response (CR) Rate
Description: nCR plus CR rate after 8 cycles of therapy as defined by the modified European Society for Bone and Marrow Transplantation (EBMT) criteria per investigator assessment as the proportion of participants with nCR or CR as their best overall response.
Time Frame: after 24 weeks (8 cycles; cycle = 21 days)
Population: Full Analysis Set (FAS): The Full analysis set (FAS) comprised of all subjects who took at least one dose of any study treatment component.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
Percentage of participants | 48.4 [33.6 to 63.2]
Statistical Analysis 1: Comparison: LBH589 + Bortezomib + Dexamethasone; Test type: Superiority; p < 0.0001, single-sample binomial test

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as time from first dose of study treatment to progression or death due to any cause, based on modified European Society for Bone and Marrow Transplantation (EBMT) criteria per Investigator's assessment
Time Frame: duration of study up to approx. 4 years
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
months | 15.3 [10.4 to 31.4]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants with CR, nCR or partial response (PR) based on modified EBMT criteria per investigator assessment
Time Frame: 24 weeks (8 cycles; cycle = 21 days)
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
Percentage of participants | 80.6 [62.5 to 92.5]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from first dose of study treatment to death
Time Frame: up to 30 days after end of study, approx. 4 years
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
months | NA [NA to NA] — N/A = not estimable as most of the participants were still alive and censored.

5. Secondary Outcome: Minimal Response Rate (MRR) Per Investigator
Description: MRR is based on modified EBMT criteria per investigator assessment
Time Frame: after 24 weeks (8 cycles; cycle = 21 days)
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
Percentage of participants | 9.7

6. Secondary Outcome: Time to Response (TTR) Per Investigator
Description: TTR is defined as the time from the date of first dose of study treatment to first documented response (PR or nCR or CR) per modified EBMT criteria as assessed by investigator
Time Frame: duration of study up to approx. 4 years
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
months | 1.4 [0.7 to 2.1]

7. Secondary Outcome: Time to Progression/Relapse (TTP) Per Investigator
Description: TTP is defined as the time from the date of the first dose of study treatment to the date of the first documented disease progression or relapse
Time Frame: duration of study up to approx. 4 years
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
months | 15.3 [10.4 to 31.4]

8. Secondary Outcome: Duration of Response (DOR) Per Investigator
Description: DOR is defined as the time from date of the first documented CR/nCR or PR to the date of the first documented progression or relapse or death due to MM
Time Frame: duration of study up to approx. 4 years
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
months | 22.7 [9.7 to 30.5]

9. Secondary Outcome: Quality of Life (QoL) as Measured by FACT/GOG-Ntx Total Score
Description: QoL as measured by Functional Assessment of Cancer Therapy/ Gynecology Oncology Group Neurotoxicity (FACT/GOG-NTX) scale calculated scores and changes from baseline were summarized by visit. The FACT/GOG-Ntx is a measure to assess neurotoxicity from systemic chemotherapy. The recall period for this measure is the past 7 days. FACT/GOG-Ntx Total Score: 0 - 152 (28 + 28 + 24 + 28 + 44 = 152). (FACT-G Physical Well-Being Score: 0 - 28, FACT-G Social/Family Well-Being Score: 0 - 28, FACT-G Emotional Well-Being Score: 0 - 24, FACT-G Functional Well-Being Score: 0 - 28, FACT/GOG-Ntx Neurotoxicity Subscale Score: 0 - 44). 4. The scales are combined. The higher the score, the better the QOL.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, and 156
Population: FAS: The FAS comprised of all subjects who took at least one dose of any study treatment component.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 31
scores on a scale
  Baseline | 112.33 [80.7 to 144.5]
  Week 12: number analyzed (Participants) | 22
  Week 12 | 91.75 [65.7 to 147.0]
  Week 24: number analyzed (Participants) | 17
  Week 24 | 100.33 [59.2 to 149.0]
  Week 36: number analyzed (Participants) | 7
  Week 36 | 125.83 [91.0 to 149.0]
  Week 48: number analyzed (Participants) | 6
  Week 48 | 114.25 [101.7 to 145.0]
  Week 60: number analyzed (Participants) | 2
  Week 60 | 109.92 [82.5 to 137.3]
  Week 72: number analyzed (Participants) | 1
  Week 72 | 108.00 [108.0 to 108.0]
  Week 84: number analyzed (Participants) | 2
  Week 84 | 101.00 [92.0 to 110.0]
  Week 96: number analyzed (Participants) | 3
  Week 96 | 121.67 [86.5 to 133.0]
  Week 108: number analyzed (Participants) | 2
  Week 108 | 120.17 [117.0 to 123.3]
  Week 120: number analyzed (Participants) | 2
  Week 120 | 125.25 [124.7 to 125.8]
  Week 132: number analyzed (Participants) | 2
  Week 132 | 114.00 [109.3 to 118.7]
  Week 156: number analyzed (Participants) | 1
  Week 156 | 119.8 [119.8 to 119.8]

10. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: AUClast, AUC0-24h, AUC0-48h, AUCinf
Description: PK sample collection was performed in subjects who agreed to blood samplings for the PK assessments of PAN and BTZ. The order of administration of the 3 study treatment components was 1) PAN, 2) Dex, and 3) BTZ.
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h, 48h post dose
Population: PAS: Pharmacokinetic Analysis Set (PAS): The PK analysis set for PAN (PAS-PAN) consisted of all subjects with at least one evaluable PK concentration of PAN. The PK analysis set for BTZ (PAS-BTZ) consisted of all subjects with at least one evaluable PK concentration of BTZ.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
h.ng/mL
  PAN: AUClast C1D1 | 106 (14.7)
  PAN: AUClast C1D8: number analyzed (Participants) | 7
  PAN: AUClast C1D8 | 156 (31.7)
  BJB432: AUClast C1D1 | 37.8 (38.2)
  BJB432: AUClast C1D8: number analyzed (Participants) | 7
  BJB432: AUClast C1D8 | 166 (87.7)
  PAN: AUC0-24h C1D1 | 87.1 (13.7)
  PAN: AUC0-24h C1D8: number analyzed (Participants) | 7
  PAN: AUC0-24h C1D8 | 125 (30.1)
  BJB432: AUC0-24h C1D1 | 18.5 (33.9)
  BJB432: AUC0-24h C1D8: number analyzed (Participants) | 7
  BJB432: AUC0-24h C1D8 | 83.8 (76.1)
  PAN: AUC0-48h C1D1 | 106 (14.8)
  PAN: AUC0-48h C1D8: number analyzed (Participants) | 7
  PAN: AUC0-48h C1D8 | 156 (31.7)
  BJB432: AUC0-48h C1D1: number analyzed (Participants) | 7
  BJB432: AUC0-48h C1D1 | 36.8 (40.6)
  BJB432: AUC0-48h C1D8: number analyzed (Participants) | 6
  BJB432: AUC0-48h C1D8 | 169 (98.8)
  PAN: AUCinf C1D1 | 116 (15.5)
  PAN: AUCinf C1D8: number analyzed (Participants) | 7
  PAN: AUCinf C1D8 | 175 (32.7)
  BJB432: AUCinf C1D1: number analyzed (Participants) | 0
  BJB432: AUCinf C1D8: number analyzed (Participants) | 0

11. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: Cmax
Description: Cmax: The maximum (peak) observed plasma concentration. PK sample collection was performed in subjects who agreed to blood samplings for the PK assessments of PAN and BTZ. The order of administration of the 3 study treatment components was 1) PAN, 2) Dex, and 3) BTZ.
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h, 48h post dose
Population: Pharmacokinetic Analysis Set (PAS): The PK analysis set for PAN (PAS-PAN) consisted of all subjects with at least one evaluable PK concentration of PAN. The PK analysis set for BTZ (PAS-BTZ) consisted of all subjects with at least one evaluable PK concentration of BTZ.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
ng/mL
  PAN: Cycle 1 Day 1 (C1D1) | 11.5 (30.4)
  PAN: Cycle 1 Day 8 (C1D8): number analyzed (Participants) | 7
  PAN: Cycle 1 Day 8 (C1D8) | 18.2 (41.5)
  BJB432: C1D1 | 1.06 (42.1)
  BJB432: C1D8: number analyzed (Participants) | 7
  BJB432: C1D8 | 4.38 (84.2)

12. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: Tmax
Description: Tmax: The time to reach maximum (peak) plasma concentration. PK sample collection was performed in subjects who agreed to blood samplings for the PK assessments of PAN and BTZ. The order of administration of the 3 study treatment components was 1) PAN, 2) Dex, and 3) BTZ.
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h, 48h post dose
Population: as for outcome 10
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
hour (h)
  PAN: C1D1 | 2.00 [1.00 to 4.00]
  PAN: C1D8: number analyzed (Participants) | 7
  PAN: C1D8 | 2.00 [0.533 to 3.08]
  BJB432: C1D1 | 24.0 [4.00 to 48.0]
  BJB432: C1D8: number analyzed (Participants) | 7
  BJB432: C1D8 | 24.0 [3.00 to 24.1]

13. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: T1/2
Description: T1/2: The elimination half-life associated with the terminal slope (Lambda_z) of a semi logarithmic concentration-time curve
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h 48h post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
hour (h)
  PAN: C1D1 | 13.7 (21.7)
  PAN: C1D8: number analyzed (Participants) | 7
  PAN: C1D8 | 16.5 (5.2)
  BJB432: C1D1: number analyzed (Participants) | 0
  BJB432: C1D8: number analyzed (Participants) | 0

14. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: Lambda_z
Description: Lambda_z: The terminal elimination rate constant (h-1)
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h 48h post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
1/hour (1/h)
  PAN: C1D1 | 0.0506 (21.7)
  PAN: C1D8: number analyzed (Participants) | 7
  PAN: C1D8 | 0.0421 (5.2)
  BJB432: C1D1: number analyzed (Participants) | 0
  BJB432: C1D8: number analyzed (Participants) | 0

15. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: CL/F
Description: CL/F: The apparent total body clearance of drug from the plasma
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h 48h post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/hour (L/h)
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
Litre/hour (L/h)
  PAN: C1D1 | 172 (15.5)
  PAN: C1D8: number analyzed (Participants) | 7
  PAN: C1D8 | 114 (32.7)
  BJB432: C1D1: number analyzed (Participants) | 0
  BJB432: C1D8: number analyzed (Participants) | 0

16. Secondary Outcome: Composite PharmacoKinetics (PK) of Panobinostat and Bortezomib: Vz/F
Description: Vz/F: The apparent volume of distribution during terminal phase (associated with Lambda_z)
Time Frame: Predose, 0.5h, 1h, 2h, 3h, 4h 8h, 24h 48h post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | LBH589 + Bortezomib + Dexamethasone
Number analyzed (Participants) | 8
Litre (L)
  PAN: C1D1 | 3390 (20.2)
  PAN: C1D8: number analyzed (Participants) | 7
  PAN: C1D8 | 2720 (31.6)
  BJB432: C1D1: number analyzed (Participants) | 0
  BJB432: C1D8: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 985 days on panobinostat + bortezomib + dexamethasone (PAN + BTZ + Dex).
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus 30 days post treatment.
Arm/Group | LBH589 + Bortezomib + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 14/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 + Bortezomib + Dexamethasone (N=31)
Coagulopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cataract (Eye disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Platelet count decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 + Bortezomib + Dexamethasone (N=31)
Anaemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Cataract (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 25
Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Face oedema (General disorders) | 2
Fatigue (General disorders) | 10
Injection site reaction (General disorders) | 3
Malaise (General disorders) | 10
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 7
Hepatic function abnormal (Hepatobiliary disorders) | 4
Conjunctivitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 3
C-reactive protein increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 9
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 7
Neuropathy peripheral (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5
Somnolence (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 7
Pollakiuria (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02290431/SAP_000.pdf
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT02290431/Prot_001.pdf